CLINICAL TRIAL: NCT03019497
Title: Towards Optimization of Traumatic Cognitive-behavioral Therapy for Treatment of Post-traumatic Stress Disorder and Related Problems
Brief Title: Cognitive-behavioral Therapy for Treatment of Post-traumatic Stress Disorder and Related Problems
Acronym: CBT-PTSD-RP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal (Other)
Responsible Party: Principal Investigator, Stephane Guay, Professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 365935
Record Dates: First submitted 2017-01-09; First posted 2017-01-12 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: PTSD
Keywords: PTSD; Related Problems; Therapy; Traumatic Event; Quality of Life; Cognitive Behavioral Therapy (CBT); Major depression; Sleep disorders; Pain; Stressors; Social support; Substance use disorder; Anxiety disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Sleep Wake Disorders; Pain; Substance-Related Disorders; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT-E (Experimental): CBT-E refers to Cognitive Behavioral Therapy with specific modules. In the CBT-E condition and following the identification of the needs identified during the evaluation, additional strategies will be added to the CBT strategies for PTSD to address one or more of the seven related problem types that emerged as a result of the traumatic event: 1) major depression, 2) sleep disorders, 3) pain, 4) stressors, 5) inadequate social support, 6) substance use disorder, and 7) anxiety disorder.
  Interventions: Behavioral: Specific Modules; Behavioral: Cognitive behavioral therapy
- CBT-C (Active Comparator): CBT-C refers to Cognitive Behavioral Therapy without specific modules. CBT-C participants will be offered only cognitive-behavioral intervention strategies to alleviate the symptoms of each of the PTSD diagnostic criteria.
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Specific Modules — Educational session about a specific related problem
  Arms: CBT-E
Behavioral: Cognitive behavioral therapy — PTSD of participants in both conditions will be addressed with cognitive-behavioral intervention strategies. These strategies are: (a) psychoeducation on PTSD, (b) anxiety management training, (c) restructuring irrational thoughts, (d) imaginative and / or in vivo exposure to memories and situations avoided, and (e) strategies for the prevention of relapse.

SUMMARY:
The purpose of this study is to evaluate the efficacy of a form of cognitive behavioral therapy (CBT) in a population of individuals with PTSD and common related problems (depression, anxiety or sleep disorders, pain, psychosocial stressors, low social support, substance use disorder). Half of the participants will receive a cognitive behavioral therapy with specific modules for the treatment of related problems (CBT-E) and the other half of participants will receive therapy without specific modules (CBT-C).

The main assumption is that participants treated in the CBT-E condition will present a lower level of symptom intensity of PTSD and a higher remission rate than those in the CBT-C condition during the post-treatment assessment. As a secondary objective, an analysis of the different parameters of effectiveness of the two forms of CBT (e.g., average number of sessions required to reach remission, treatment strategies used) will be performed.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) will affect nearly one in ten Canadians in their lifetime and more than 75% of them will develop at least one other related problem (i.e. depression). Results from a previous study suggest that CBT offering a flexible number of sessions and support for common related problems can improve the effectiveness of CBT. However, no studies have demonstrated the superior efficacy of flexible CBT compared to CBT targeting only PTSD to individuals with PTSD and common related problems.

A randomized parallel-stratified single-blind controlled trial will be used. Randomization will be performed through www.randomized.net, a comprehensive internet-based randomization service for clinical trials, with multiple Coordinating Center users (each with their own role). A total of 134 individuals will be randomized to one of two therapy conditions. Following the initial assessment, between 8 and 32 sessions with a psychologist will be offered to participants upon achievement of remission of the diagnosis of PTSD. Discontinuation of treatment will be decided in collaboration with the participant and will be considered on the basis of achieving a non-clinical severity level of symptoms of PTSD on the PCL-5 (i.e., score <33 and absence or non-clinical level of severity of each of the symptoms). The participants will be re-evaluated 3 times after their therapy (1 week, 3 months and 6 months post-therapy) on primary and secondary measures. A 1 year post-therapy follow-up will also be provided for the primary measure only.

Planned analysis. The statistical analysis will respect the "intent-to-treat" principle: the results of all randomized participants will be included in the groups in which they were originally assigned. The significance level is fixed at .05 and bilateral tests will be used. With regards to missing data, first the type of missing data will be determined (e.g. missing completely randomly). Thereafter, a multiple imputation strategy (3 to 5 imputations) will be used to replace the data and carry out the various analysis planned. This data replacement strategy is recognized as being robust and efficient in addition to resolving uncertainty due to missing data. Generalized linear models will be used to execute group comparisons (CBT-C vs CBT-E) on the main measurements using the pre-treatment (T0) result as a covariate. The same strategy will be used for comparisons of the secondary variables and related problems. An analysis of the different parameters of effectiveness of the two forms of CBT (e.g. average number of sessions required to achieve remission, treatment strategy used) will be carried out.

Subgroup analysis. No subgroup analysis is expected. Exploratory analysis will be conducted to determine if the results are generalizable to victims of both sexes and to the two major categories of traumatic exposures characterizing the sample recruited, namely violent criminal acts and workplace accidents.

Sample size and calculations of treatment effects. Based on the treatment effect size observed in a pilot study on the effects of CBT-E, similar research, and on the use of the GPower power calculation software, the sample size required to obtain statistical power of .80 with 3 follow-ups, a significance level at .05 and bilateral testing for ANCOVA is 53 participants per group. A sample of 106 participants will allow for detections of differences in means between the two groups in terms of symptoms intensity of PTSD. It will also be adequate to verify the other assumptions and objectives of this project. Based on data from our recent studies on the efficacy of CBT-C, and the literature on similar therapies (Bradley et al., 2005), the attrition rate is estimated to be 28% for participants who will be randomized in CBT-C. For CBT-E, the attrition rate observed during a pilot project was 14% (3 dropouts out of 21 participants). Given these attrition rates, recruitment for each of the therapies to achieve the required statistical power is calculated as follows: CBT-C = 53 participants * attrition (28%) = 74; CBT-E = 53 participants * attrition (14%) = 60). Consequently, a total of 134 participants will be randomized to one of the two conditions of therapy.

Selection bias: The assignment to the intervention will be made only after the participant has agreed to participate in the study. Bias in statistical analysis: In order to minimize biases, the analysis will be carried out in a single-blind manner, the statistician will not know which intervention refers to the code assigned to each of them in the database. Bias resulting from missing data and dropouts: All analysis will follow the "intent to treat" principle, in order to minimize biases stemming from missing data and drop-outs during the intervention.

Conducting a clinical trial on comparing the effectiveness of CBT with or without specific modules for patients with PTSD and related problems will increase the efficacy of CBT, innovate in the delivery of CBT, and improve the training of current and future clinicians. The results could also encourage victims' compensation boards to adjust their practices and thus improve the health of the beneficiaries.

ELIGIBILITY:
Inclusion Criteria:

* Exposed to a traumatic event at an adult age
* Primary PTSD diagnosis according to the DSM-5 criteria
* At least one PTSD related problem (depressive, anxiety or sleep disorders, pain, psychosocial stressors, inadequate social support, substance use disorder)
* Being fluent in French.

Exclusion Criteria:

* Schizophrenia diagnostic, current or past psychotic episodes, bipolar disorder, organic cerebral disorder or intellectual deficiency
* Presence of a trouble linked to a substance developed prior to the traumatic event
* Physical condition preventing participation in the study (e.g. cerebral trauma)
* Presence of active suicide ideas.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5; Weathers et al., 2013) | Baseline, changes from baseline at 1 week post-treatment, 3 months post-treatment, and 6 months post-treatment
  The CAPS-5 will be used to evaluate the presence 20 symptoms indicative of PTSD according to the DSM-5. This scale was designed not only to assess symptoms but also to provide indications regarding symptoms onset and duration, associated subjective distress, perceived impact of symptoms on social and professional functioning, changes in symptomology since the previous CAPS assessment and global severity of PTSD.

SECONDARY OUTCOMES:
The Structured Clinical Interview (SCID-I; First, Spitzer, Gibbon & Williams, 1995) | Baseline, 1 week post-treatment, 3 months post-treatment, 6 months post-treatment
  SCID-I will be used to evaluate the presence of Axis-1 disorders other than acute stress disorder according to the DSM-5.
The Beck II Depression Inventory (BDI-II; Beck, Steer & Brown, 1996) | Baseline, 1 week post-treatment, 3 months post-treatment, 6 months post-treatment
  BDI-II consists of 21 items intended to assess the presence and severity of depressive symptoms in the last two weeks.
The Beck Anxiety Inventory (BAI; Beck, Epstein, Brown & Steer, 1988) | Baseline, 1 week post-treatment, 3 months post-treatment, 6 months post-treatment
  BAI is a self-reported 21-item instrument assessing the main symptoms experienced by clinically anxious individuals as defined by the DSM-IV. Participants rate the intensity of symptoms experienced over the past week on a scale ranging from 0 (Not al all) to 3 (A lot).
The WHOQOL - Bref (WHOQOL Group, 1998) | Baseline, every 4 weeks during treatment, 1 week post-treatment, 3 months post-treatment, 6 months post-treatment, 1 year post-treatment
  WHOQOL is a 26 items self-reported measure that will be used to evaluate the quality of life in four key spheres of life: physical health, quality of the environment, mental health and social relations.
The Inventory of Social Support in Anxious Situations (ISSAS; St-Jean-Trudel et al., 2005) | Baseline, 1 week post-treatment, 3 months post-treatment, 6 months post-treatment
  ISSAS will be used to evaluate the frequency of different types of supporting behaviors and the perception thereof in anxiety-provoking situations.The questionnaire contains 31 items divided in two dimensions, negative and positive social support.
The Pittsburgh Sleep Quality Index (PSQI) | Baseline, 1 week post-treatment, 3 months post-treatment, 6 months post-treatment
  PSQI is a self-report questionnaire containing 19 items evaluating seven components of sleep quality: (a) subjective quality of sleep; (b) sleep latency; (c) sleep duration; (d) sleep efficiency; (e) sleep perturbation; (f) intake of hypnotic medications and (g) impact on daily activities. A scale ranging from 0 to 3 is used to measure each component; the sum of which provides researchers with a global indication of sleep quality on a scale ranging from 0 to 21. An addendum of seven additional items targeting sleep difficulties specific to individuals suffering from PTSD will also be used and has been previously validated (Germain, Hall, Krakow, Shear, & Buysse, 2005).
The Life Events Questionnaire (LEQ; Norbeck, 1984) | Baseline, 1 week post-treatment, 3 months post-treatment, 6 months post-treatment
  LEQ is an 82-item self-report questionnaire that will be used to evaluate the presence of potentially stressful life events over a determined period. The instrument has 9 dimensions (e.g. parenthood, justice) and participants must determine if the event had a positive or negative impact on their life before quantifying the severity of this impact (none, low, average, important).
The Brief Pain Inventory (BPI; Cleeland, 1989) | Baseline, 1 week post-treatment, 3 months post-treatment, 6 months post-treatment
  BPI will be used to evaluate the pain severity and its interference. The sub-scale assessing pain severity has 4 items, each using a Likert scale ranging from 0 (no pain) to 10 (the worst pain you can imagine). The second sub-scale, evaluating pain interference, contains 7 items, each using Likert scale ranging from 0 (no interference) to 10 (interferes severely).
The Health Cost Interview | Baseline, 3 months post-treatment
  The Health Cost Interview is a semi-structured interview comprising of 19 items. It has been used previously by other researchers (Roberge, Marchand, Reinharz, Marchand, & Cloutier, 2004; Roberge et al., 2005; Poirier-Bisson et al., 2013) to determine the costs associated with healthcare service use as well as costs attributed to absenteeism and work-related sick leaves since the traumatic event. The interview includes items on the consultations with medical professionals, both generalists and specialists, as well as with allied health professionals (e.g. psychologist, social worker). It also assesses the medication intake and work absenteeism.
The Social Provisions Scale (SPS; Cutrona & Russel, 1987) | Baseline, 1 week post-treatment, 3 months post-treatment, 6 months post-treatment
  SPS will be used to evaluate the perceptions regarding social support in general. This 24-item questionnaire measures six dimensions of social support: 1) emotional support, 2) tangible and material help, 3) advice, 4) social integration, 5) self-esteem and 6) the need to feel useful and needed.
The Posttraumatic Stress Disorder Checklist Scale-version DSM-5 (PCL-5; Weathers, Litz et al., 2013) | Baseline, changes from baseline at every 4-sessions during treatment (i.e. session 4, 8 … 28 - the number of assessments during treatment will vary based on the number of sessions), 1 week, 3 months, 6 months and 1 year post-treatment.
  PCL-5 will be used as a follow-up measure to assess PTSD symptoms in the last month according to the DSM-5.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Guay, PhD, Principal Investigator — Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal
Locations (1):
- Stephane Guay, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradley R, Greene J, Russ E, Dutra L, Westen D. A multidimensional meta-analysis of psychotherapy for PTSD. Am J Psychiatry. 2005 Feb;162(2):214-27. doi: 10.1176/appi.ajp.162.2.214. PMID 15677582
- [Background] Blake DD, Weathers FW, Nagy LM, Kaloupek DG, Gusman FD, Charney DS, Keane TM. The development of a Clinician-Administered PTSD Scale. J Trauma Stress. 1995 Jan;8(1):75-90. doi: 10.1007/BF02105408. PMID 7712061
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Poirier-Bisson J, Marchand A, Pelland ME, Lessard MJ, Dupuis G, Fleet R, Roberge P. Incremental cost-effectiveness of pharmacotherapy and two brief cognitive-behavioral therapies compared with usual care for panic disorder and noncardiac chest pain. J Nerv Ment Dis. 2013 Sep;201(9):753-9. doi: 10.1097/NMD.0b013e3182a2127d. PMID 23995030
- [Background] Galovski TE, Blain LM, Mott JM, Elwood L, Houle T. Manualized therapy for PTSD: flexing the structure of cognitive processing therapy. J Consult Clin Psychol. 2012 Dec;80(6):968-81. doi: 10.1037/a0030600. Epub 2012 Oct 29. PMID 23106761
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Norbeck JS. Modification of life event questionnaires for use with female respondents. Res Nurs Health. 1984 Mar;7(1):61-71. doi: 10.1002/nur.4770070110. PMID 6565302
- [Background] Roberge P, Marchand A, Reinharz D, Cloutier K, Mainguy N, Miller JM, Begin J, Turcotte J. Healthcare utilization following cognitive-behavioral treatment for panic disorder with agoraphobia. Cogn Behav Ther. 2005;34(2):79-88. doi: 10.1080/16506070510008443. PMID 15986784
- [Background] Roberge P, Marchand A, Reinharz D, Marchand L, Cloutier K. Évaluation économique de la thérapie cognitive-comportementale des troubles anxieux. Canadian Psychology. 2004 Aug;45(3):202-216.
- [Background] St-Jean-Trudel E, Guay S, Marchand A, O'Connor K. [Elaboration and validation of a questionnaire measuring social support in situations of anxiety with a population of university students]. Sante Ment Que. 2005 Autumn;30(2):43-60. doi: 10.7202/012138ar. French. PMID 16505924
- [Background] Cleeland CS. (1989). Measurement of pain by subjective report. In CR Chapman and JD Loeser (eds.), Issues in pain measurement, Advances in pain research and therapy (vol. 12, p. 391-403). New York : Raven Press.
- [Background] Cutrona CE, Russell DW. The provisions of social support and adaptation to stress. Advance in Personal Relationship. 1987;(1):37-67.
- [Background] Weathers FW, Litz BT, Keane, TM, Palmieri PA, Marx BP, Schnurr, PP. The PTSD Checklist for DSM5 (PCL5). 2003; Retrieved from URL www.ptsd.va.gov.
- [Background] Beck A, Steer R, Brown G. Manuel de l'inventaire de presentation de Beck (2nd ed.). 1996; Toronto : Harcourt Brace & Company Canada.
- [Background] First MB, Williams JBW, Karg RS, Spitzer RL. User's Guide for the Structured Clinical Interview for DSM-5 Disorders, Research Version (SCID-5-RV). 2015; Arlington, VA : American Psychiatric Association.
- [Derived] O'Doherty L, Whelan M, Carter GJ, Brown K, Tarzia L, Hegarty K, Feder G, Brown SJ. Psychosocial interventions for survivors of rape and sexual assault experienced during adulthood. Cochrane Database Syst Rev. 2023 Oct 5;10(10):CD013456. doi: 10.1002/14651858.CD013456.pub2. PMID 37795783